CLINICAL TRIAL: NCT05992922
Title: A Phase 2, Single-Center, Randomized, Double- Masked, Placebo-Controlled Study to Assess the Safety and Efficacy of IC265 Ophthalmic Solution 1% in Subjects Diagnosed With Dry Eye Disease
Brief Title: A Study to Assess the Safety and Efficacy of IC265 Ophthalmic Solution for Dry Eye in Adult Participants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unexpected adverse events were observed in a subset of patients on drug. In an over abundance of caution the study was terminated. All adverse events resolved with no sequelae.
Sponsor: Iacta Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-110-0002
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-09

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IC265 Ophthalmic Solution 1% (Experimental): 1 drop will be instilled in each eye twice daily.
  Interventions: Drug: IC265 Ophthalmic Solution 1%
- Placebo Ophthalmic Solution (Vehicle) (Placebo Comparator): 1 drop will be instilled in each eye twice daily.
  Interventions: Drug: Placebo Ophthalmic Solution (Vehicle)

INTERVENTIONS:
Drug: IC265 Ophthalmic Solution 1% — 1 drop will be instilled in each eye twice a day
  Arms: IC265 Ophthalmic Solution 1%
Drug: Placebo Ophthalmic Solution (Vehicle) — 1 drop will be instilled in each eye twice a day
  Arms: Placebo Ophthalmic Solution (Vehicle)

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of IC265 compared to vehicle in participants with signs and symptoms dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent
* Have a reported or documented history of dry eye for at least 6 months prior to Visit 1
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1
* Report a score of ≥ 2 on a Ocular Discomfort & 4-symptom questionnaire in at least one symptom at Visits 1 and 2
* Have a Schirmer's Test score of ≤10mm and ≥1mm in at least one eye at Visits 1and 2
* Have a pre-CAE(controlled adverse environment) (conjunctival redness score ≥ 1 according to the Conjunctival Redness for Dry Eye Scale in at least one eye at Visits 1 and 2
* Have a corneal fluorescein staining score of ≥ 2 in at least one region (e.g. inferior, superior, or central) at Visits 1 and 2
* Have a sum corneal fluorescein staining score of ≥ 4, based on the sum of the inferior, superior, and central regions at Visits 1 and 2
* Have a total lissamine green conjunctival score of ≥ 2, based on the sum of the temporal and nasal regions at Visits 1 and 2
* Demonstrate a response to the CAE at Visits 1 and 2 as defined by:

  1. Having at least a ≥1 point increase in fluorescein staining in the inferior region in at least one eye following CAE exposure
  2. Reporting an Ocular Discomfort Score ≥3 at 2 or more consecutive time points in at least one eye during CAE exposure (if a subject has an ocular discomfort rating of 3 at time = 0 for an eye, s/he must report an ocular discomfort rating of 4 for two consecutive measurements for that eye) Note: a subject cannot have an ocular discomfort score of 4 at time = 0)

Exclusion Criteria:

* Have any clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction, ocular rosacea, lid margin inflammation or active ocular allergies that require therapeutic treatment
* Have any clinically significant (CS) posterior chamber findings, or a history of such findings/disorders, that may include exudative (i.e., wet) age-related macular degeneration, retinal vein occlusion, diabetic retinopathy, glaucoma, ocular hypertension, or any other retinal or optic nerve disease/disorder that require therapeutic treatment and/or in the opinion of the Investigator may interfere with study parameters
* Have worn contact lenses within 48 hours prior to Visit 1 or anticipate using contact lenses during the study
* Have laser-assisted in situ keratomileusis (LASIK) or similar type of corneal refractive surgery and/or any other ocular surgical procedure within 12 months prior to Visit 1; or have any ocular surgical procedure scheduled to be conducted during the study period
* Have had any surgeries of the ocular surface or lid in the past 6 months
* Have a history of lacrimal duct obstruction in either eye within 12 months prior to Visit 1
* Have used temporary (i.e., collagen) punctal plugs within 12 weeks prior to Visit 1 or anticipate their use during the study period
* Have permanent punctal plugs inserted or removed - including falling out - or have had surgical punctal occlusion within 12 weeks prior to Visit 1 or anticipate any such event at any time during the study period
* Use any of the following treatments in the period indicated before Visit 1 or anticipate their use at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Iacta Selected Site, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
Started | 20; 20 eyes | 20; 20 eyes
Completed | 0; 0 eyes | 0; 0 eyes
Not Completed | 20; 20 eyes | 20; 20 eyes
Not completed — Adverse Event | 6 | 0
Not completed — Sponsor Termination of Study | 14 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.48) | 65.8 (11.5) | 67.1 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ocular Discomfort and Dry Eye Symptoms
Description: Subjects will rate the severity of each of the following symptoms, with regard to how both their eyes feel, in general - overall ocular discomfort, burning, dryness, grittiness and stinging according to the following 6-point (0 to 5) scale where 0 = none and 5 = worst.
Time Frame: Change from Baseline Post-CAE® (controlled adverse environment) Day 15
Population: Intent to Treat - only 14 participants in the IC265 Ophthalmic Solution 1% and 19 in the Placebo Ophthalmic Solution reached Day 15.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 14 | 19
Number analyzed (eyes) | 14 | 19
score on a scale
  Overall Ocular Discomfort | -0.6 (1.09) | 0.3 (0.82)
  Burning | -0.5 (1.34) | -0.7 (1.38)
  Dryness | -0.7 (1.27) | 0.3 (0.56)
  Grittiness | -0.4 (1.22) | 0.2 (1.38)
  Stinging | -0.8 (1.63) | -0.1 (1.15)

2. Other Pre Specified Outcome: Tear Film Break-up Time (TFBUT)
Description: With the aid of a slit-lamp, the examiner will monitor the integrity of the tear film, noting the time it takes to form micelles from the time that the eye is opened. TFBUT will be measured in seconds using a stopwatch and a digital image recording system for the right eye followed by the left eye. For each eye, 2 measurements will be taken and averaged unless the 2 measurements are > 2 seconds apart and are each < 10 seconds, in which case, a third measurement would be taken and the 2 closest of the 3 would be averaged.
Time Frame: Change from Baseline Pre-CAE® (controlled adverse environment) in TFBUT in Study Eye Day 15
Population: Change from Baseline Pre-CAE® in TFBUT in Study Eye - Intent-to-Treat Population. Only 14 participants in the IC265 Ophthalmic Solution 1% and 19 in the Placebo Ophthalmic Solution reached Day 15.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 14 | 19
Number analyzed (eyes) | 14 | 19
seconds | 1.357 (0.5310) | 0.883 (0.4572)

3. Other Pre Specified Outcome: Ocular Surface Disease Index (OSDI)©
Description: Change from baseline to Visit 3 (Day 15). Subjects will complete the OSDI© questionnaire. The OSDI© is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease. the OSDI© is a valid and reliable instrument for measure dry eye disease (normal, mild to moderate, and severe) and effects vision-related function.
Time Frame: Day 15
Population: Only 14 participants in the IC265 Ophthalmic Solution 1% and 19 in the Placebo Ophthalmic Solution reached Day 15.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 14 | 19
Number analyzed (eyes) | 14 | 19
score on a scale | -3.0 (15.45) | -0.5 (12.12)

4. Other Pre Specified Outcome: Schirmer's Test
Description: Change from Baseline. Schirmer Tear Test will be performed according to the following procedure:
  * Using a sterile Tear Flo Schirmer test strip, a bend in the strip will be made in line with the notch in the strip.
  * The subject will be instructed to gaze up and in.
  * The Schirmer test strip will be placed in the lower temporal lid margin of each eye such that the strip fits tightly. Subjects will be instructed to close their eyes.
  * After 5 minutes have elapsed, the Schirmer strip will be removed. The length of the moistened area will be recorded (mm) for each eye.
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 14 | 19
Number analyzed (eyes) | 14 | 19
mm | 0.57 (3.567) | 1.95 (8.721)

5. Other Pre Specified Outcome: Ocular Discomfort During CAE - Change From Baseline to Visit 3
Description: Change from Baseline in Ora to Visit 3 Calibra® Ocular Discomfort Scale During the CAE® in the Study Eye. Ocular discomfort scores will be subjectively graded by the subjects according to the following scale: 0 - no discomfort, 1 - intermittent awareness, 2 - constant awareness, 3 - intermittent discomfort, 4 - constant discomfort.
Time Frame: Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 14 | 19
Number analyzed (eyes) | 14 | 19
score on a scale
  0 Minutes | -0.4 (0.84) | 0.2 (0.60)
  5 Minutes | -0.1 (0.73) | -0.1 (0.85)
  10 Minutes | -0.1 (0.66) | -0.2 (0.83)
  15 Minutes | 0.1 (1.00) | 0.1 (0.71)
  20 Minutes | -0.1 (0.86) | 0.1 (0.62)
  25 Minutes | -0.1 (0.73) | 0.1 (0.97)
  30 Minutes | -0.3 (0.73) | 0.0 (0.75)
  35 Minutes | -0.2 (0.80) | 0.1 (0.85)
  40 Minutes | -0.1 (0.77) | 0.1 (0.66)
  45 Minutes | -0.1 (0.77) | 0.2 (0.60)
  50 Minutes | -0.1 (0.77) | 0.2 (0.60)
  55 Minutes | -0.1 (0.77) | 0.2 (0.63)
  60 Minutes | 0.0 (0.55) | 0.4 (0.68)
  65 Minutes | -0.1 (0.47) | 0.2 (0.71)
  70 Minutes | 0.0 (0.55) | 0.1 (0.71)
  75 Minutes | 0.0 (0.55) | 0.2 (0.69)
  80 Minutes | 0.1 (0.47) | 0.2 (0.96)
  85 Minutes | 0.0 (0.39) | 0.1 (0.78)
  90 Minutes | 0.0 (0.39) | 0.1 (0.52)

6. Other Pre Specified Outcome: Daily Diary Symptom Score
Description: Subject Daily Diary in the Evening - Day 8 to Day 14 average, Subjects will rate the severity of each of the following symptoms, with regard to how both their eyes feel, in general - overall ocular discomfort, burning, dryness, grittiness and stinging according to the following 6-point (0 to 5) scale where 0 = none and 5 = worst.The average of the daily diary scores will be summarized using continuous descriptive statistics for the time period.
Time Frame: Daily Diary Evening - Day 8 to Day 14
Population: Intent to Treat - Only 14 participants in the IC265 Ophthalmic Solution 1% and 19 in the Placebo Ophthalmic Solution provided daily diaries in this timeframe.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 14 | 19
score on a scale
  Ocular Discomfort | 2.6 (1.30) | 2.2 (1.06)
  Burning | 1.3 (1.2) | 1.5 (1.28)
  Dryness | 2.7 (1.21) | 2.6 (0.99)
  Grittiness | 2.1 (1.45) | 1.2 (1.24)
  Stinging | 1.3 (1.25) | 1.3 (1.38)

7. Other Pre Specified Outcome: Conjunctival Redness
Description: Conjunctival Redness 5 point scale (0 - Normal, without vasodilation, 1 - Trace ciliary or conjunctival vasodilation, 2 - Broad ciliary vasodilation, 3 - Broad ciliary and slight, horizontal conjunctival vasodilation, 4 - Broad ciliary and prominent, horizontal conjunctival vasodilation)
Time Frame: Change from Baseline to Day 15
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 14 | 19
Number analyzed (eyes) | 14 | 19
score on a scale | -0.3 (15.45) | -0.15 (12.12)

8. Other Pre Specified Outcome: Lissamine Green Staining in the Following Regions: Central, Superior, Inferior, Temporal, Nasal, Corneal Sum, Conjunctival Sum, and Total Eye Score
Description: Change from Baseline Pre-CAE® in Corneal Lissamine Green Staining in Study Eye. The staining will be graded with a Corneal and Conjunctival Staining Scale. The scale is a 5 point scale from 0 (no staining) to 4 (confluent).
Time Frame: Day 15
Population: Intent-to-Treat Population - Only 14 participants in the IC265 Ophthalmic Solution 1% and 19 in the Placebo Ophthalmic Solution provided daily diaries in this timeframe.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 14 | 19
Number analyzed (eyes) | 14 | 19
score on a scale
  Inferior | 0.50 (0.920) | 0.32 (1.017)
  Superior | 0.43 (1.107) | 0.55 (0.985)
  Central | 0.43 (0.756) | 0.32 (0.582)
  Temporal | -0.07 (0.616) | -0.05 (0.864)
  Nasal | 0.07 (0.584) | 0.11 (0.658)
  Corneal Sum | 1.36 (2.089) | 1.18 (2.129)
  Conjunctival Sum | 0.00 (0.941) | 0.05 (1.177)
  Total Sum | 1.36 (2.825) | 1.24 (2.791)

9. Other Pre Specified Outcome: Fluorescein Staining in the Following Regions: Central, Superior, Inferior, Temporal, Nasal, Corneal Sum, Conjunctival Sum, and Total Eye Score
Description: Change from Baseline Pre-CAE® to Post-CAE® in Corneal Fluorescein Staining in the Study Eye. The staining will be graded with a Corneal and Conjunctival Staining Scale. The scale is a 5 point scale from 0 (no staining) to 4 (confluent).
Time Frame: Day 15
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
Number analyzed (Participants) | 14 | 19
Number analyzed (eyes) | 14 | 19
score on a scale
  Inferior | -0.32 (0.750) | -0.55 (0.832)
  Superior | -0.21 (0.752) | 0.26 (1.046)
  Central | -0.04 (1.308) | 0.24 (1.147)
  Temporal | 0.07 (0.675) | 0.39 (0.809)
  Nasal | 0.11 (0.836) | -0.08 (0.886)
  Corneal Sum | -0.57 (2.165) | -0.05 (2.598)
  Conjunctival Sum | 0.18 (0.868) | 0.32 (1.406)
  Total Sum | -0.39 (2.558) | 0.26 (3.048)

ADVERSE EVENTS:
Time Frame: The adverse events were collected over the duration of the trial out to Visit 3, Day 15. The study was terminated early and patients were discontinued from study drug.
Arm/Group | IC265 Ophthalmic Solution 1% | Placebo Ophthalmic Solution (Vehicle)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 20/20 | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC265 Ophthalmic Solution 1% (N=20) | Placebo Ophthalmic Solution (Vehicle) (N=20)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC265 Ophthalmic Solution 1% (N=20) | Placebo Ophthalmic Solution (Vehicle) (N=20)
Corneal neovascularisation (Eye disorders) | 0 (0) | 1 (1)
Corneal Opacity (Eye disorders) | 11 (11) | 0 (0)
Eye Pruritus (Eye disorders) | 2 (2) | 0 (0)
Instillation site foreign body sensation (Eye disorders) | 1 (1) | 0 (0)
Instillation site irritation (Eye disorders) | 15 (16) | 2 (2)
Lacrimation Increased (Eye disorders) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 5 (5) | 1 (1)
Visual Acuity reduced (Eye disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early, Visit 3 Day 15, due to the unexpected epithelial haze findings in several subjects on IC265. All but one AEs of epithelial haze observed in several of subjects in IC265 OS 1% were mild and resolved without intervention in all cases. The study was discontinued in the abundance of caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT05992922/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT05992922/SAP_001.pdf